CLINICAL TRIAL: NCT02779166
Title: Evaluation of Perioperative Celecoxib for Hip Arthroscopy
Acronym: Celecoxib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Michael Terry, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00067550
Record Dates: First submitted 2016-05-13; First posted 2016-05-20 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Hip Labral Tears
Keywords: hip arthroscopy
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Received 400mg celecoxib prior to surgery
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Received placebo pill prior to surgery
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Celecoxib — Received 400mg celecoxib prior to surgery
  Arms: Intervention
Drug: placebo
  Arms: Placebo

SUMMARY:
Celecoxib is commonly used for perioperative pain control for certain orthopaedic procedures. It has been shown to be successful in assisting in pain control for knee arthroscopy. It has not previously been studied in hip arthroscopy. This is a double blinded randomized controlled trial to determine the efficacy of celecoxib in perioperative pain control for hip arthroscopy.

DETAILED DESCRIPTION:
This study examines the efficacy of perioperative dose of celecoxib in pain management after hip arthroscopy. Perioperative administration of celecoxib has been shown to improve pain control after knee arthroscopy, but this has not yet been studied in the hip. In this study, patients are randomized to receive either 400mg celecoxib or placebo 1 hour prior to undergoing hip arthroscopy surgery. Postoperatively, patients are monitored for pain on the VAS scale, narcotic use, and meeting discharge criteria. The study will enroll 100 patients. Patients are approached for informed consent on the day of surgery. Pain scores, narcotic use, and time to discharge in the celecoxib group are compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are undergoing a hip arthroscopy procedure at Northwestern Memorial Hospital with Dr. Michael Terry.

Exclusion Criteria:

* Pregnant women and any patient under the age of 18 years.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-08; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Terry, MD, Principal Investigator — Northwestern University

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: 50 patients received 400mg celecoxib prior to surgery
  Celecoxib: Received 400mg celecoxib prior to surgery
- Placebo: 48 received placebo pill prior to surgery
  placebo
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 50 | 48
Completed | 50 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Received placebo pill prior to surgery
  placebo
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 50 | 48 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 48 | 98
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (11.9) | 35.8 (11.6) | 35.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 24 | 19 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 48 | 98

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Score for Pain (VAS) in the Immediate Post Operative Period
Description: The pain VAS is a uni dimensional measure of pain intensity. It is a continuous scale comprised of a 0-10 pain rating. A score of 0 indicates no pain while a score of 10 would indicate extreme pain.
Time Frame: Pre operative on day of surgery, immediately following OR close, 1 hr post operatively, 2 hrs post operatively
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 50 | 48
score on a scale
  Pre-Operative VAS Score | 2.11 (2.06) | 2.33 (1.98)
  Immediate Post Op VAS Score | 4.41 (3.00) | 5.02 (3.10)
  1 hr Post Op VAS Score | 4.63 (1.91) | 5.36 (1.92)
  2 hr Post Op VAS Score | 4.11 (1.75) | 4.92 (1.98)

2. Primary Outcome: Total Narcotic Consumption in the Post Anesthesia Care Unit (PACU)
Description: Monitored consumption of narcotic medications following surgery, measured in morphine equivalents
Time Frame: duration of PACU stay,immediate post op period up to a maximum of 4 hours postoperatively
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 50 | 48
morphine milligram equivalents | 15.326 (11.0) | 15.419 (13.2)

3. Primary Outcome: Time to Discharge Following Surgery
Description: Total time to discharge from OR close following surgery, measured in minutes
Time Frame: time from OR to discharge, up to a maximum of 6 hours postoperatively
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 50 | 48
minutes | 152.9 (55.2) | 172.9 (57.6)

ADVERSE EVENTS:
Arm/Group | Intervention | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/48
Other Adverse Events (participants affected / at risk) | 0/50 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No